CLINICAL TRIAL: NCT03003143
Title: Effect of Vigabatrin in Refractory Autoimmune Encephalitis Patients - A Pilot Study
Brief Title: Effect of Vigabatrin in Refractory Autoimmune Encephalitis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1607092776
Record Dates: First submitted 2016-12-13; First posted 2016-12-26 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Autoimmune Encephalopathy
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Vigabatrin

ARMS (1):
- Vigabatrin treatment group (Experimental)
  Interventions: Drug: Vigabatrin 500 MG

INTERVENTIONS:
Drug: Vigabatrin 500 MG

SUMMARY:
Investigation of efficacy of vigabatrin in refractory autoimmune encephalitis patients

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Possible autoimmune encephalitis
* Patients who have been diagnosed and treated for encephalitis for more than 4 weeks
* Patients with epilepsy (EEG finding or clinically)

Exclusion Criteria:

* septic shock, fever >38.5 ℃, O2 saturation <90%, respiratory rate >25, HR >120
* previously, mRS=3 or mRS>3
* MMSE<20
* Patients who have terminal disease
* eye problem
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Seizure frequency reduction | 3 month of vigabatrin administration
  50% reduction - favorable outcome

SECONDARY OUTCOMES:
Modified Rankin Scale | 3 month of vigabatrin administration
Quality of life (Quality of Life in Epilepsy Inventory, QOLIE-31) | after 3 month of vigabatrin administration
Depression (Beck Depression Inventory®-II) | 3 month of vigabatrin administration
Cognition (Mini-Mental State Examination-Korean) | 3 month of vigabatrin administration
Sleep quality (Pittsburgh Sleep Quality Assessment) | 3 month of vigabatrin administration

CONTACTS AND LOCATIONS:
Overall Officials: KON CHU, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Bjurstom H, Wang J, Ericsson I, Bengtsson M, Liu Y, Kumar-Mendu S, Issazadeh-Navikas S, Birnir B. GABA, a natural immunomodulator of T lymphocytes. J Neuroimmunol. 2008 Dec 15;205(1-2):44-50. doi: 10.1016/j.jneuroim.2008.08.017. Epub 2008 Oct 26. PMID 18954912
- [Background] Rossi S, Muzio L, De Chiara V, Grasselli G, Musella A, Musumeci G, Mandolesi G, De Ceglia R, Maida S, Biffi E, Pedrocchi A, Menegon A, Bernardi G, Furlan R, Martino G, Centonze D. Impaired striatal GABA transmission in experimental autoimmune encephalomyelitis. Brain Behav Immun. 2011 Jul;25(5):947-56. doi: 10.1016/j.bbi.2010.10.004. Epub 2010 Oct 20. PMID 20940040